CLINICAL TRIAL: NCT00175019
Title: A Phase 3, Open-Label, Randomized, Allopurinol-Controlled Study to Assess the Long-Term Safety of Oral Febuxostat in Subjects With Gout
Brief Title: Allopurinol Versus Febuxostat in Subjects Completing the Phase 3 Trials C02-009 or C02-010
Acronym: EXCEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C02-021; U1111-1113-9814 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Gout
Keywords: uric acid; xanthine oxidase; hyperuricemia; tophi; Drug Therapy
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Febuxostat 80 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Febuxostat 120 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Allopurinol QD (Active Comparator)
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Febuxostat — Febuxostat 80 mg, tablets, orally, once daily.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 80 mg QD
Drug: Febuxostat — Febuxostat 120 mg, tablets, orally, once daily.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 120 mg QD
Drug: Allopurinol — Allopurinol 100 mg or 300 mg, tablets, orally, once daily.
  Other Names: Zyloprim
  Arms: Allopurinol QD

SUMMARY:
The purpose of this study is to determine the long-term safety of febuxostat, once daily (QD), compared to allopurinol in reducing serum urate levels in subjects with gout.

DETAILED DESCRIPTION:
Uric acid is the end product of purine degradation in humans. Hyperuricemia, a urate concentration in serum exceeding the limit of urate solubility (approximately 7.0 mg/dL), is a common biochemical abnormality. Aberrations in any of the multiple mechanisms involved in the production and/or excretion of uric acid may increase serum urate concentrations, with persistent hyperuricemia as a marker for extracellular fluid monosodium urate supersaturation. As such, hyperuricemia is a necessary (but often insufficient) risk factor for monosodium urate crystal deposition in tissues and is the fundamental pathophysiological process underlying the clinical manifestations of gout, which is a chronic disease characterized by urate crystal formation and deposition in joints and bones. Gout may progress from episodic attacks of acute inflammatory arthritis to a disabling chronic disorder characterized by deforming arthropathy; destructive deposits of urate crystals (tophi) in bones, joints, and other organs; structural and functional renal impairment due to interstitial urate crystal deposition; and urinary tract stones composed entirely or partially of uric acid crystals. Management of gout requires chronic treatment aimed at lowering serum urate levels into a subsaturating range (usually <6.0 mg/dL) in which crystal formation and deposition are prevented or reversed.

Febuxostat (TMX-67) is a non-purine selective xanthine oxidase inhibitor being developed as an orally administered agent for the management of hyperuricemia in patients with gout.

This study was originally designed and initiated having all subjects initially assigned to 80 mg febuxostat provided as an 80 mg tablet, to be administered orally. Subjects could be titrated to 120 mg, provided as one 40 and 80 mg tablet, between Months 2 and 6, if their serum uric acid rose > 6.0 mg/dL; the dose could be down-titrated to 80 mg if the serum uric acid decreased to < 3.0 mg/dL.

The protocol was amended to add a comparator arm, and to have subjects randomized to 80 or 120 mg febuxostat or allopurinol (100 or 300 mg, dependent on renal function). The information below reflects the treatments following the implementation of the revised protocol.

ELIGIBILITY:
Inclusion Criteria:

* Is receiving thiazide diuretic therapy (only to subjects randomized to or receiving febuxostat).
* Has a serum urate level less than 8.0 mg/dL and is not taking uric acid-lowering therapy (other than allopurinol or febuxostat).
* Has participated in a clinical study in which febuxostat was administered.
* Is completing Phase 3 Studies C02-009 or C02-010.
* Must not have experienced any serious study drug-related adverse events in the previous study.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study

Exclusion Criteria:

* Has had any other significant medical condition as defined by the investigator that would interfere with the treatment, safety, or compliance with the protocol.
* Is intolerant of allopurinol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1086 (Actual)
Dates: Start 2003-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda

REFERENCES:
- [Result] Becker MA, Schumacher HR, MacDonald PA, Lloyd E, Lademacher C. Clinical efficacy and safety of successful longterm urate lowering with febuxostat or allopurinol in subjects with gout. J Rheumatol. 2009 Jun;36(6):1273-82. doi: 10.3899/jrheum.080814. Epub 2009 Mar 13. PMID 19286847
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 174 investigative sites, including 168 in the United States and 6 in Canada, from 28 July 2003 to 26 February 2007.
Pre-assignment Details: Subjects were to have completed either 28 weeks or 52 weeks of double-blind dosing in Study C02-009 (NCT00174915) or C02-010 (NCT00102440), respectively before enrollment.
Groups:
- Febuxostat 80 mg QD: Febuxostat 80 mg, taken orally, once daily.
- Febuxostat 120 mg QD: Febuxostat 120 mg, taken orally, once daily
- Allopurinol QD: Allopurinol 100 mg or 300 mg, tablets, orally, once daily.
Period: Overall Study
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Started | 606 (Based on final stable treatment in C02-021, defined as after dose switch not allowed.) | 388 (Based on final stable treatment in C02-021, defined as after dose switch not allowed.) | 92 (Based on final stable treatment in C02-021, defined as after dose switch not allowed.)
Completed | 412 (Based on final stable treatment in C02-021, defined as after dose switch not allowed.) | 217 (Based on final stable treatment in C02-021, defined as after dose switch not allowed.) | 35 (Based on final stable treatment in C02-021, defined as after dose switch not allowed.)
Not Completed | 194 | 171 | 57
Not completed — Adverse Event | 54 | 22 | 2
Not completed — Protocol Violation | 6 | 3 | 3
Not completed — Lost to Follow-up | 42 | 39 | 9
Not completed — Did not continue under Amendment 4 | 1 | 1 | 2
Not completed — Personal Reason(s) | 39 | 31 | 8
Not completed — Therapeutic Failure | 10 | 38 | 22
Not completed — Gout Flare | 2 | 3 | 0
Not completed — Reason Not Specified | 40 | 34 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD | Total
Number analyzed (Participants) | 606 | 388 | 92 | 1086
Age Continuous [Mean (Standard Deviation); unit: years] — Based on Final Stable Treatment in study C02-021
  years | 53.0 (11.74) | 48.4 (11.02) | 51.3 (12.72) | 51.2 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Based on Final Stable Treatment in study C02-021
  Participants
    Female | 25 | 17 | 2 | 44
    Male | 581 | 371 | 90 | 1042
Presence of Tophus [Number; unit: participants] — Based on Final Stable Treatment in study C02-021
  participants
    Present | 116 | 83 | 15 | 214
    Absent | 490 | 305 | 77 | 872
Race/Ethnicity [Number; unit: participants] — Based on Final Stable Treatment in study C02-021
  participants
    Asian | 15 | 9 | 4 | 28
    Black or African American | 47 | 33 | 16 | 96
    White | 499 | 299 | 64 | 862
    Hispanic | 30 | 29 | 7 | 66
    Other | 15 | 18 | 1 | 34
Renal Function [Number; unit: participants] — Based on Final Stable Treatment in study C02-021. Impaired defined as serum creatinine <1.5 mg/dL.
  participants
    Normal | 593 | 381 | 92 | 1066
    Impaired | 13 | 7 | 0 | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Based on Final Stable Treatment in study C02-021
  kg/m² | 31.9 (5.49) | 34.1 (6.71) | 32.4 (5.58) | 31.9 (5.49)
Serum Urate [Mean (Standard Deviation); unit: mg/dL] — Based on Final Stable Treatment in study C02-021
  mg/dL | 9.65 (1.20) | 10.05 (1.29) | 9.83 (1.27) | 9.81 (1.25)

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline to the Last Visit on Treatment.
Description: The percent change in serum urate from baseline to the last visit on treatment was summarized. The last visit on treatment was the last visit at which a serum urate value was collected prior to any changes in drug and/or dose from the initial treatment assignment.
Time Frame: Last Visit on treatment (up to 40 months).
Population: Results were summarized by the initial treatment the subject was assigned to before any changes in drug and/or dose. All subjects with a post-baseline serum urate level measurement while receiving their initial treatment were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 636 | 283 | 141
percent change from baseline | -46.69 (17.43) | -52.99 (19.12) | -32.17 (17.71)

2. Secondary Outcome: Percent Change From Baseline in Primary Tophus Size at Month 12 for Subjects With Palpable Tophi Measured at Baseline.
Description: The area of the primary tophus was calculated based on the length and width of the tophus measured at the Month 12 visit. The percent change from baseline in primary tophus size to the Month 12 visit was summarized.
Time Frame: Month 12
Population: Results were summarized by final stable treatment which was the treatment a subject was receiving after drug and/or dose changes were no longer allowed. Subjects with a primary tophus at baseline which was also measured at the Month 12 visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 80 | 51 | 9
percent change from baseline | -82 [-100 to -40] | -79 [-100 to -26] | -56 [-100 to -16]

3. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to < 6.0 mg/dL at Month 1.
Description: Serum urate values were obtained at the Month 1 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 1 visit was summarized.
Time Frame: Month 1
Population: Results were summarized by the initial treatment the subject was assigned to before any changes in drug and/or dose. Subjects with a serum urate value at the Month 1 visit and who had not changed from their initial treatment were included in the analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 620 | 277 | 139
percentage of subjects | 80.8 | 87.0 | 46.0

4. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to < 6.0 mg/dL at Month 12.
Description: Serum urate values were obtained at the Month 12 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 12 visit was summarized.
Time Frame: Month 12
Population: Results were summarized by the initial treatment the subject was assigned to before any changes in drug and/or dose. Subjects with a serum urate value at the Month 12 visit and who had not changed from their initial treatment were included in the analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 422 | 168 | 45
percentage of subjects | 88.9 | 86.3 | 82.2

5. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to < 6.0 mg/dL at Month 24.
Description: Serum urate values were obtained at the Month 24 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 24 visit was summarized.
Time Frame: Month 24
Population: Results were summarized by the initial treatment the subject was assigned to before any changes in drug and/or dose. Subjects with a serum urate value at the Month 24 visit and who had not changed from their initial treatment were included in the analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 364 | 141 | 42
percentage of subjects | 89.3 | 87.2 | 78.6

6. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to < 6.0 mg/dL at Month 36.
Description: Serum urate values were obtained at the Month 36 visit. The percentage of subjects whose serum urate was <6.0 mg/dL at the Month 36 visit was summarized.
Time Frame: Month 36
Population: Results were summarized by the initial treatment the subject was assigned to before any changes in drug and/or dose. Subjects with a serum urate value at the Month 36 visit and who had not changed from their initial treatment were included in the analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 120 | 47 | 10
percentage of subjects | 90.8 | 91.5 | 90.0

7. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreases to < 6.0 mg/dL at Last Visit on Treatment.
Description: The percentage of subjects whose serum urate was <6.0 mg/dL at the last visit on treatment was summarized. The last visit on treatment was the last visit at which a serum urate value was collected prior to any changes in drug and/or dose from the initial treatment assignment.
Time Frame: Last Visit on treatment (up to 40 months).
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 636 | 283 | 141
percentage of subjects | 70.8 | 82.0 | 32.6

8. Secondary Outcome: Percent Change From Baseline in Primary Tophus Size at Month 24 for Subjects With Palpable Tophi Measured at Baseline.
Description: The area of the primary tophus was calculated based on the length and width of the tophus measured at baseline and Month 24 visit. The percent change from baseline in primary tophus size to the Month 24 visit was summarized.
Time Frame: Month 24
Population: Results were summarized by final stable treatment which was the treatment a subject was receiving after drug and/or dose changes were no longer allowed. Subjects with a primary tophus at baseline which was also measured at the Month 24 visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 64 | 32 | 4
percent change from baseline | -100 [-100 to -54] | -96 [-100 to -52] | -87 [-98 to -29]

9. Secondary Outcome: Percent Change From Baseline in Primary Tophus Size at Month 36 for Subjects With Palpable Tophi Measured at Baseline.
Description: The area of the primary tophus was calculated based on the length and width of the tophus measured at baseline and Month 36 visit. The percent change from baseline in primary tophus size to the Month 36 visit was summarized.
Time Frame: Month 36
Population: Results were summarized by final stable treatment which was the treatment a subject was receiving after drug and/or dose changes were no longer allowed. Subjects with a primary tophus at baseline which was also measured at the Month 36 visit were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 1 | 0 | 0
percent change from baseline | -83 [-83 to -83] |  |

10. Secondary Outcome: Percent Change From Baseline in Primary Tophus Size at Final Visit for Subjects With Palpable Tophi Measured at Baseline.
Description: The area of the primary tophus was calculated based on the length and width of the tophus measured at baseline and final visit. The percent change from baseline in primary tophus size to the final visit was summarized.
Time Frame: Final Visit (up to 40 months).
Population: Results were summarized by final stable treatment which was the treatment a subject was receiving after drug and/or dose changes were no longer allowed. Subjects with a primary tophus at baseline which was also measured while receiving their final stable treatment were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 107 | 76 | 14
percent change from baseline | -96 [-100 to -42] | -84 [-100 to -16] | -67 [-100 to 0]

11. Secondary Outcome: Percent Change From Baseline in the Total Number of Tophi for Subjects With Palpable Tophi at Final Visit.
Description: The number of tophi were counted at baseline and final visits. The percent change from baseline in the number of tophi to the final visit was summarized.
Time Frame: Final Visit (up to 40 months).
Population: Results were summarized by final stable treatment which was the treatment a subject was receiving after drug and/or dose changes were no longer allowed. Subjects with a primary tophus at baseline who also had their tophi counted while receiving their final stable treatment were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 107 | 76 | 14
percent change from baseline | -59.9 (45.9) | -58.3 (42.5) | -48.7 (42.5)

12. Secondary Outcome: Percentage of Subjects Requiring Treatment for Gout Flare up to Month 12.
Description: The percentage of subjects requiring treatment for gout flare during the first twelve months of final stable treatment was summarized.
Time Frame: Month 12
Population: Results were summarized by final stable treatment which was the treatment a subject was receiving after drug and/or dose changes were no longer allowed. A subject who reported more than one gout flare during the time interval was counted only once.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 606 | 388 | 92
percentage of subjects | 29.4 | 42.5 | 28.3

13. Secondary Outcome: Percentage of Subjects Requiring Treatment for Gout Flare After Month 12.
Description: The percentage of subjects requiring treatment for gout flare after the first 12 months of final stable treatment was summarized.
Time Frame: After Month 12 to Final Visit
Population: as for outcome 12
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Number analyzed (Participants) | 516 | 293 | 56
percentage of subjects | 15.3 | 19.8 | 23.2

ADVERSE EVENTS:
Arm/Group | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Allopurinol QD
Serious Adverse Events (participants affected / at risk) | 98/801 | 50/487 | 16/178
Other Adverse Events (participants affected / at risk) | 444/801 | 257/487 | 66/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 80 mg QD (N=801) | Febuxostat 120 mg QD (N=487) | Allopurinol QD (N=178)
Anaemia Deficiencies (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenias (Blood and lymphatic system disorders) | 1 | 0 | 0
Aortic Valvular Disorders (Cardiac disorders) | 1 | 0 | 0
Cardiac Conduction Disorders (Cardiac disorders) | 2 | 0 | 0
Cardiomyopathies (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disorders not elsewhere classified (NEC) (Cardiac disorders) | 13 | 6 | 1
Heart Failures NEC (Cardiac disorders) | 3 | 3 | 1
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 17 | 3 | 2
Myocardial Disorders NEC (Cardiac disorders) | 1 | 0 | 0
Supraventricular Arrhythmias (Cardiac disorders) | 1 | 2 | 1
Ventricular Arrhythmias and Cardiac Arrest (Cardiac disorders) | 2 | 0 | 0
Male Reproductive Tract Disorders Congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hearing Losses (Ear and labyrinth disorders) | 0 | 1 | 0
Inner Ear Signs and Symptoms (Ear and labyrinth disorders) | 0 | 2 | 0
Abdominal Hernias, Site Unspecified (Gastrointestinal disorders) | 0 | 2 | 0
Benign Neoplasms GastrointestinaI (Excluding Oral Cavity) (Gastrointestinal disorders) | 1 | 2 | 0
Colitis (Excluding Infective) (Gastrointestinal disorders) | 1 | 1 | 0
Diaphragmatic Hernias (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal and Small Intestinal Stenosis and Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Atonic and Hypomotility Disorders NEC (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Disorders NEC (General disorders) | 1 | 0 | 0
Gastrointestinal Stenosis and Obstruction NEC (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernias (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Ulcers and Perforation NEC (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical Hernias (Gastrointestinal disorders) | 0 | 0 | 1
Hernias NEC (General disorders) | 1 | 0 | 0
Pain and Discomfort NEC (General disorders) | 1 | 2 | 0
Bile Duct Infections and Inflammations (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis and Cholelithiasis (Hepatobiliary disorders) | 7 | 1 | 1
Hepatocellular Damage and Hepatitis NEC (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal and Gastrointestinal Infections (Infections and infestations) | 3 | 2 | 2
Bacterial Infections NEC (Infections and infestations) | 3 | 1 | 0
Bone and Joint Infections (Infections and infestations) | 1 | 0 | 0
Cardiac Infections (Infections and infestations) | 1 | 0 | 0
Infections NEC (Infections and infestations) | 5 | 0 | 0
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 7 | 2 | 0
Sepsis, Bacteraemia, Viraemia, and Fungaemia NEC (Infections and infestations) | 3 | 0 | 0
Staphylococcal Infections (Infections and infestations) | 2 | 0 | 0
Upper Respiratory Tract Infections (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infections (Infections and infestations) | 1 | 0 | 0
Cardiac and Vascular Procedural Complications (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cerebral Injuries NEC (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injuries NEC (Including Traumatic Amputation) (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb Fractures and Dislocations (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle, Tendon and Ligament Injuries (Injury, poisoning and procedural complications) | 1 | 1 | 0
Non-Site Specific Injuries NEC (Injury, poisoning and procedural complications) | 4 | 0 | 0
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 4 | 0 | 0
Neurologic Diagnostic Procedures (Investigations) | 1 | 0 | 0
Diabetes Mellitus (Including Subtypes) (Metabolism and nutrition disorders) | 0 | 1 | 0
General Nutritional Disorders NEC (Metabolism and nutrition disorders) | 0 | 1 | 0
Magnesium Metabolism Disorders (Metabolism and nutrition disorders) | 1 | 0 | 0
Potassium Imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Bone Disorders NEC (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral Disc Disorders (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Joint Related Disorders NEC (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle Related Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Spine and Neck Deformities (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
B-cell Lymphomas NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bile Duct Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast and Nipple Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colonic Neoplasms Malignant (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Endocrine Neoplasms Benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasms Benign Site Unspecified NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-Small Cell Malignant/Respiratory Tract Cell Type Specified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian Neoplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic Neoplasms Malignant (Excl Islet Cell and Carcinoid) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Central Nervous System Haemorrhages and CVA (Nervous system disorders) | 6 | 2 | 0
Central Nervous System Vascular Disorders NEC (Nervous system disorders) | 2 | 1 | 0
Cervical Spinal Cord and Nerve Root Disorders (Nervous system disorders) | 0 | 0 | 1
Disturbances in Consciousness NEC (Nervous system disorders) | 2 | 2 | 0
Neurologic Visual Problems NEC (Nervous system disorders) | 0 | 0 | 1
Neurological Signs and Symptoms NEC (Nervous system disorders) | 1 | 0 | 0
Paralysis and Paresis (Excl Cranial Nerve) (Nervous system disorders) | 1 | 0 | 0
Transient Cerebrovascular Events (Nervous system disorders) | 0 | 1 | 0
Renal Failure and Impairment (Renal and urinary disorders) | 3 | 0 | 0
Renal Lithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal Vascular and Ischaemic Conditions (Psychiatric disorders) | 0 | 1 | 0
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bronchospasms and Obstruction (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Lower Respiratory Tract Inflam. and Immunologic Conditions (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Thrombotic and Embolic Conditions (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Apocrine and Eccrine Gland Disorders (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Neoplasms Benign (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic Aneurysms and Dissections (Vascular disorders) | 2 | 1 | 0
Non-Site Specific Necrosis and Vascular Insufficiency NEC (Vascular disorders) | 1 | 0 | 0
Peripheral Aneurysms and Dissections (Vascular disorders) | 0 | 1 | 0
Peripheral Embolism and Thrombosis (Vascular disorders) | 2 | 0 | 1
Peripheral Vascular Disorders NEC (Vascular disorders) | 2 | 0 | 0
Peripheral Vasoconstriction, Necrosis and Vascular Insuff. (Vascular disorders) | 1 | 0 | 0
Vascular Hypertensive Disorders NEC (Vascular disorders) | 2 | 0 | 1
Vascular Hypotensive Disorders NEC (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 80 mg QD (N=801) | Febuxostat 120 mg QD (N=487) | Allopurinol QD (N=178)
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 38 | 33 | 4
Oedema NEC (General disorders) | 49 | 17 | 3
Influenza Viral Infections (Infections and infestations) | 44 | 16 | 2
Lower Respiratory Tract and Lung Infections (Infections and infestations) | 60 | 27 | 6
Upper Respiratory Tract Infections (Infections and infestations) | 246 | 119 | 30
Joint Related Signs and Symptoms (Musculoskeletal and connective tissue disorders) | 100 | 50 | 12
Musculoskeletal and Connective Tissues Signs and Symptoms NEC (Musculoskeletal and connective tissue disorders) | 140 | 82 | 23
Headache NEC (Nervous system disorders) | 45 | 38 | 7
Dermatitis and Eczema (Skin and subcutaneous tissue disorders) | 44 | 23 | 2
Vascular Hypertensive Disorders NEC (Vascular disorders) | 67 | 41 | 5

LIMITATIONS AND CAVEATS:
Subjects may receive >1 treatment. Adverse events are summarized by treatment at time of observation and subjects who receive >1 treatment are summarized for each treatment they receive, so subjects at risk will not match number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.